CLINICAL TRIAL: NCT02458664
Title: BASE HSP110 : A New Therapeutic Target and a New Marker for Prognosis of Type MSI Colorectal Cancer
Acronym: BASE HSP110
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: NI12029; 2013-A01080-45 (Other Grant/Funding Number: N° ID RCB)
Record Dates: First submitted 2015-05-27; First posted 2015-06-01 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Rectum Cancer; Cancer of Colon
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colo-rectal cancer: All patients undergoing curative colorectal cancer in general and digestive surgery department at Saint-Antoine hospital
  Interventions: Genetic: Genetic analysis on tumor kept in tumor bank

INTERVENTIONS:
Genetic: Genetic analysis on tumor kept in tumor bank

SUMMARY:
We collect prospectively and retrospectively, patients' demographic, pathological, surgical, therapeutic and prognosis informations in a database. After patient's consent to collect tumoural samples of their colorectal cancer after resection.

We will then be able to evaluate the impact of HSP110, a chaperon protein, on their prognosis. Other proteins (to be determined) will also be study, after.

DETAILED DESCRIPTION:
To investigate the importance of HSP110DE9 as a prognostic marker for colorectal cancer, we will analyze genotyping fluorescence quantitative RT-PCR and / or immunomarquage the presence of this mutant in a large cohort of patients (more than 2000 patients had or having a colorectal cancer). All patients have been or will be made in general and digestive surgery department at Saint-Antoine hospital. Tumor fragments samples were or will be made on their tumor and keep it in the tumor bank of the Saint-Antoine hospital. All patients reported their no objection to the use of these tumor fragments for research purposes. A database will be built and correlated with the tumor fragments. This project is intended that the constitution of a clinical database including prognostic so that we make discoveries on HSP110DE9 or other molecular biology to discover markers can be correlated with clinical data. In the absence of other studies on the subject, with no real knowledge of the prognostic impact of this mutant, we cannot provide an effective computation. We therefore propose to make a database of 2000 patients retrospectively and prospectively to obtain statistical results valid and powerful.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing curative colorectal cancer in general and digestive surgery department at Saint-Antoine hospital.
* Patients reporting their non-opposition to the use of tissue samples taken from their specimen for research purposes.

Exclusion Criteria:

* Patients who did not report their non-opposition to the use of tissue samples taken from their specimen for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, male or female, over 18 years, undergoing curative colorectal resection
Sampling Method: Non-Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2013-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival and Recurrence free survival after resection of the colon cancer | End of follow up : at least 3 years
  3 years for prospective patients, more for retrospective patients

SECONDARY OUTCOMES:
Overall survival | End of follow up : at least 3 years
  3 years for prospective patients, more for retrospective patients

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Digestive Surgery, Hôpital Saint-Antoine, Paris, France, France